CLINICAL TRIAL: NCT02631109
Title: L-DEP Regimen as a Salvage Therapy for Refractory Epstein Barr Virus-induced Hemophagocytic Lymphohistiocytosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Doctor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-DEP-EBV-HLH
Record Dates: First submitted 2015-12-03; First posted 2015-12-16 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Pegaspargase; hemophagocytic lymphohistiocytosis; Epstein Barr virus
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Epstein-Barr Virus Infections | interventions — pegaspargase; Doxorubicin; Etoposide; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-DEP (Experimental): Pegaspargase 2000U/m2 day5; doxorubicin (doxorubicin hydrochloride liposome injection) 25 mg/m2 day 1; etoposide 100 mg/m2 was administered once on the first day of every week; methylprednisolone 15 mg/kg days 1 to 3, 0.75 mg/kg days 4 to 7
  Interventions: Drug: Pegaspargase; Drug: doxorubicin; Drug: etoposide; Drug: methylprednisolone

INTERVENTIONS:
Drug: Pegaspargase — 2000U/m2 day5
Drug: doxorubicin — 25mg/m2 day1
Drug: etoposide — 100 mg/m2 was administered once on the first day of every week
Drug: methylprednisolone — 15 mg/kg days 1 to 3, 0.75 mg/kg days 4 to 7

SUMMARY:
This study aimed to investigate the efficacy and safety of Pegaspargase together with liposomal doxorubicin, etoposide and high dose methylprednisolone (L-DEP) as a salvage therapy for refractory Epstein Barr virus-induced hemophagocytic lymphohistiocytosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were older than 14 years of age
2. Diagnosed as EBV-Hemophagocytic Lymphohistiocytosis (HLH)
3. Patients did not achieve at lease partial response after initial treatment including HLH-94 or DEP no less than 2 weeks
4. Informed consent

Exclusion Criteria:

1. Heart function above grade II (NYHA)
2. Accumulated dose of doxorubicin above 300mg/m2 or epirubicin above 450mg/m2
3. Pregnancy or lactating Women
4. Allergic to Pegaspargase, doxorubicin or etoposide
5. Active bleeding of the internal organs
6. uncontrollable infection
7. history of acute and chronic pancreatitis
8. Participate in other clinical research at the same time

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment response | Change from before and 2,4,6 and 8 weeks after initiating L-DEP salvage therapy
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT).
  A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5× 109/L; for patients with a neutrophil count of 0.5 to 2.0 × 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT decrease of at least 50%.
Change of Epstein-Barr virus(EBV)-DNA | Change from before and 2, 4, 6 and 8 weeks after initiating L-DEP salvage therapy

SECONDARY OUTCOMES:
Survival | from the time patients received L-DEP salvage therapy up to 24 months or November 2019
Adverse events that are related to treatment | through study completion, an average of 2 years
  Adverse events including pancreatitis, liver function damage, myelosuppression, infection, bleeding and so on.

CONTACTS AND LOCATIONS:
Overall Officials: zhao wang, M.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Wang Y, Huang W, Hu L, Cen X, Li L, Wang J, Shen J, Wei N, Wang Z. Multicenter study of combination DEP regimen as a salvage therapy for adult refractory hemophagocytic lymphohistiocytosis. Blood. 2015 Nov 5;126(19):2186-92. doi: 10.1182/blood-2015-05-644914. Epub 2015 Aug 19. PMID 26289641
- [Derived] Wang J, Wang Y, Wu L, Zhang J, Lai W, Wang Z. PEG-aspargase and DEP regimen combination therapy for refractory Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis. J Hematol Oncol. 2016 Sep 9;9(1):84. doi: 10.1186/s13045-016-0317-7. PMID 27613189